CLINICAL TRIAL: NCT03936517
Title: Safety and Efficacy of Prednisolone in Adrenal Insufficiency Disease (PRED-AID Study)
Acronym: PRED-AID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Imperial Health Charity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18IC4546; 2018-001502-28 (EudraCT Number); 201045 (Other: IRAS); ISRCTN41325341 (Registry Identifier: ISRCTN); 19/LO/0083 (Other: Research Ethics Committee)
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Adrenal Insufficiency
Keywords: Glucocorticoids; Hydrocortisone; Prednisolone; Cortisol
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Prednisolone; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Two-arm, two-period, double-blind randomised crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomised to one of two arms: A) prednisolone in the first treatment period and hydrocortisone in the second period; or B) hydrocortisone in the first treatment period and prednisolone in the second period.
  Blinding will be achieved by providing participants with a tablet three times a day regardless of the treatment they are currently on. If on a hydrocortisone treatment period, the participant will receive tablets of hydrocortisone at their personally tailored dose three times a day (morning, noon and afternoon). When on prednisolone, the participant will receive a prednisolone tablet in the morning (at their personal dose), followed by a matched placebo at noon and in the afternoon. The tablets used in the study have been specifically made for the study to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone first; hydrocortisone second (Other): Participant will receive 4 months of prednisolone in the first study period and 4 months of hydrocortisone in the second study period.
  Interventions: Drug: Prednisolone; Drug: Hydrocortisone
- Hydrocortisone first; prednisolone second (Other): Participant will receive 4 months of hydrocortisone in the first study period and 4 months of prednisolone in the second study period.
  Interventions: Drug: Prednisolone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Prednisolone — Low dose prednisolone for the treatment of adrenal insufficiency. Usually administered once daily
Drug: Hydrocortisone — Standard regimens of hydrocortisone for the treatment of adrenal insufficiency. Usually administered thrice daily.

SUMMARY:
This study compares low-dose prednisolone therapy against standard regimens of hydrocortisone therapy for the treatment of adrenal insufficiency (AI). AI is a condition in which, individuals are unable to sufficiently produce the natural stress hormone, cortisol.

DETAILED DESCRIPTION:
Steroid replacement therapy is vital for the health of patients with adrenal insufficiency (AI), who are unable to produce the natural stress hormone, cortisol. The objectives of steroid replacement therapy are to replace the body's physiological requirements for cortisol without over-replacement and consequent Cushing's syndrome. Equally, under-replacement presents the risk of patients experiencing potentially fatal Addisonian crises.

Appropriately replacing a patient's steroid requirement is a significant challenge. Hydrocortisone (HC) is used in the majority of patients with AI in the UK. However, HC has a short duration of action, necessitating dosing 3 times a day. Low-dose prednisolone (PR) is an alternative to HC which needs only once-daily. There have been no studies directly comparing low-dose PR to HC treatment.

This is a two-arm, two-period, double-blind, randomised, cross-over study comparing the low dose PR and standard regimens of HC in the treatment of AI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 70 years
* Male or female
* Diagnosed with AI for over 6 months according to standard diagnostic criteria
* Established on stable HC replacement or prednisolone replacement, dose not altered for at least 3 months
* Established on a stable dose of Fludrocortisone, if taking, dose not altered for at least 3 months
* Participants taking other hormone replacements (e.g. levothyroxine, testosterone or growth hormone in secondary adrenal insufficiency) are accepted providing that their replacement doses have not altered for at least 3 months
* Participants who are otherwise healthy enough to participate, as determined by pre-study medical history and physical examination.
* Participants who are able and willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Participants with a diagnosis of Type 1 or Type 2 diabetes mellitus.
* Unable to give informed consent.
* Taking supplements or herbal medications that the participant is unwilling or unable to stop prior to and during the study period e.g. St John's Wort (may decrease prednisolone levels), Cat's claw, Echinacea (immunomodulatory properties).
* Currently taking medications that alter CYP3A4 metabolism of glucocorticoids that the participant is unwilling or unable to stop prior to and during the study period e.g. phenytoin, phenobarbital, rifampicin, rifabutin, carbamazepine, primidone, aminoglutethimide, itraconazole, ketoconazole, ciclosporin or ritonavir.
* Pregnancy, taking the combined oral contraceptive pill, or oral oestrogen replacement therapy due to the effects on cortisol binding globulin levels and determination of prednisolone levels. Transdermal oestrogen replacement is permitted.
* Diagnosis of congenital adrenal hyperplasia, untreated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of Osteocalcin | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  Assesses bone health of each group by comparing total osteocalcin and undercarboxylated osterocalcin

SECONDARY OUTCOMES:
Change in concentration of P1NP | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  Assesses bone health of each group by comparing P1NP
Change in concentration of BALP | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  Assesses bone health of each group by comparing BALP
Change in concentration of NTX | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  Assesses bone health of each group by comparing NTX
Heart Rate | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  recording observations- heart rate
Systolic and diastolic blood pressure | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  recording observations- blood pressure
Waist-Hip circumference | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  recording observations- Waist-Hip circumference ratios
Change in concentration of Lipid profile (Total cholesterol, HDL, LDL and triglycerides) | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  measuring biochemical indicators of cardiovascular risk: total cholesterol, HDL, LDL and triglycerides
Change in concentration of high sensitivity CRP | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  measuring biochemical indicators of cardiovascular risk: high sensitivity CRP
Change in concentration of Glucose | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  measuring glucose
Change in concentration of HbA1c | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  measuring HbA1c
Infection rates and severity | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  assessed by completion of the German National Cohort Questionnaire (GNCQ). Frequency (None; 1; 2; 3; >3; Unknown) of 1. Upper respiratory tract infections; 2. Lower respiratory tract infections; 3.Gastroenteritis; 4. Mucosal infections; 5. Urinary tract infections; 6. Influenza; will be recorded. The frequencies of each type of infection will be compared between time points.
Wellbeing assessed by completion the short form health survey | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  assessed by completion the short form health survey-36 (SF-36). Scores will be produced in each of 8 domains (Physical functioning, Role functioning/physical, Role functioning/emotional, Energy/fatigue, Emotional wellbeing, Social functioning, Pain, General Health and Health Change). Each domain is scored from 0 to 100, with higher scores suggesting more positive outcomes. Scores will be compared in each domain between time points.
Wellbeing assessed by completion the Addi-QoL questionnaire | Between Day 1 and Day 120 within each study period; and between Day 120 of Period 1 and Period 2.
  assessed by completion the Addi-QoL questionnaire. A total score between 30 and 120 is produced, with higher scores suggesting a more positive outcome. The score is compared between time points.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Meeran, MBBS BSc MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No